CLINICAL TRIAL: NCT01266707
Title: Phase 1 Study of HLA-A*2402 Restricted Antiangiogenic Peptide Vaccine Therapy Using Epitope Peptide Derived Feom VEGFR1 and VEGFR2 in Treating Patients With Unresectable, Recurrent, or Metastatic Hepatocellular Carcinoma
Brief Title: Antiangiogenic Peptide Vaccine Therapy in Treating Patient With Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fukushima Medical University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Fukushima Medical University, Fukushima Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 560
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; peptide vaccine; VEGFR
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (Experimental): VEGRF1, VEGFR2
  Interventions: Biological: antiangiogenic paptide vaccine

INTERVENTIONS:
Biological: antiangiogenic paptide vaccine — for drugs include administration time frame
  Other Names: VEGFR1 and VEGFR2 specific epitope vaccine

SUMMARY:
The purpose of this study is to assess toxicities of angiogenic peptide vaccine therapy in treating HLA-A*2402 restricted patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
It has been required to develop new treatment modalities for patients with advanced heptatocellular carcinoma. Immunotherapy is one of the encouraging modalities for patients. We have to assess its toxicities, clinical response and immune responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or treatment-resistant patients with Hepatocellular carcinoma
* Measurable disease by CT scan
* ECOG performance status 0-2
* Life expectancy > 3 months
* Laboratory values as follows: 2,000/mm3 < WBC <15,000/mm3, Platelet counts > 75,000/mm3, Total Bilirubin < 1.5 mg/dl, Asparate transaminase < 150IU/L, Alanine transaminase < 150 IU/L, Creatinine < 3.0mg/dl
* HLA-A*2402
* Able and willing to give valid written informed consent

Exclusion Criteria:

* Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
* Brest-feeder
* Active or uncontrolled infection
* Steroids or immunosuppressing agent dependent status
* Active or uncontrolled other malignancy
* Serious or uncured wound
* Decision of unsuitableness by principal investigator or physician-in charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2007-03; Primary Completion 2012-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Toxicities as assessed by NCI-CACAE ver3 | 3 months

SECONDARY OUTCOMES:
Differences of peptide specific CTL response in vitro among sequence of peptide vaccine administration | 3 months
CD8 population | 3 months
Change in level of regulatory T cells | 3 months
Objective response rate | 1 year
Feasibility | 1 year
Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mitsukazu Gotoh, PhD & MD, Study Chair — Fukushima Medical University, Department of Regeneration Surgery
Locations (1):
- Fukushima Medical University Hospital, Fukushima, Fukushima, Japan

REFERENCES:
- [Background] Niethammer AG, Xiang R, Becker JC, Wodrich H, Pertl U, Karsten G, Eliceiri BP, Reisfeld RA. A DNA vaccine against VEGF receptor 2 prevents effective angiogenesis and inhibits tumor growth. Nat Med. 2002 Dec;8(12):1369-75. doi: 10.1038/nm1202-794. Epub 2002 Nov 4. PMID 12415261
- [Background] Ishizaki H, Tsunoda T, Wada S, Yamauchi M, Shibuya M, Tahara H. Inhibition of tumor growth with antiangiogenic cancer vaccine using epitope peptides derived from human vascular endothelial growth factor receptor 1. Clin Cancer Res. 2006 Oct 1;12(19):5841-9. doi: 10.1158/1078-0432.CCR-06-0750. PMID 17020992
- [Background] Wada S, Tsunoda T, Baba T, Primus FJ, Kuwano H, Shibuya M, Tahara H. Rationale for antiangiogenic cancer therapy with vaccination using epitope peptides derived from human vascular endothelial growth factor receptor 2. Cancer Res. 2005 Jun 1;65(11):4939-46. doi: 10.1158/0008-5472.CAN-04-3759. PMID 15930316